CLINICAL TRIAL: NCT00887978
Title: A 16-Week, International, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Oral UT-15C Sustained Release Tablets in Subjects With Pulmonary Arterial Hypertension
Brief Title: Efficacy and Safety of Oral UT-15C Tablets to Treat Pulmonary Arterial Hypertension
Acronym: FREEDOM-C2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDE-PH-308
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Identical placebo tablets to UT-15C, doses were titrated in the same manner
  Interventions: Drug: Placebo
- UT-15C SR (Experimental): Doses were initiated at 0.25 mg BID and increased by 0.25 mg BID every three days (as clinically indicated based on tolerability and symptoms of PAH), to a max dose of 16 mg BID.
  Interventions: Drug: UT-15C SR

INTERVENTIONS:
Drug: UT-15C SR — treprostinil diolamine sustained release tablets
  Other Names: treprostinil diolamine, treprostinil diethanolamine, UT-15C
  Arms: UT-15C SR
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is an international, multi-center, randomized, double-blind, placebo-controlled study in subjects with PAH who are currently receiving approved therapy for their PAH (i.e., endothelin receptor antagonist and/or phosphodiesterase-5 inhibitor). Study visits will occur at 4 week intervals for 16 weeks with the key measure of efficacy being the 6-minute walk test. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, and exercise tests.

Patients who complete all assessments for 16-weeks will also be eligible to enter an open-label, extension phase study (FREEDOM - EXT).

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible for inclusion in this study if all of the following criteria apply:
* Between 18 and 75 years of age, inclusive.
* Body weight at least 40 kg (approximately 90 lbs.)
* PAH that is either idiopathic/heritable; associated with appetite suppressant or toxin use; associated with collagen vascular disease; associated with repaired congenital shunts; associated with HIV.
* Currently receiving an approved endothelin receptor antagonist and/or an approved phosphodiesterase-5 inhibitor for at least 90 days and on a stable dose for at least the last 30 days.
* Baseline six-minute walk distance (6MWD) between 150-425 meters
* Previous testing (e.g., right heart catheterization, echocardiography) consistent with the diagnosis of PAH.
* Reliable and cooperative with protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Rubin, MD, Study Chair — University of California, San Diego
Locations (62):
- United States (40):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialist, LTD, Phoenix, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - UCSD Medical Center, La Jolla, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Florida-Jacksonville, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Pulmonary Critical Care Medicine, Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Presbyterian Medical Center, New York, New York
  - Mary M Parkes Center for Asthma, Allergy and Pulmonary Care, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Lindner Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The University of Toledo, Toledo, Ohio
  - Legacy Pulmonary Northwest, Portland, Oregon
  - OHSU, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Transplant Center, Falls Church, Virginia
- University Hospital Gasthuisberg, Leuven, Belgium
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - Vancouver Coastal Health Respiratory Clinic, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
- France (3):
  - Hospital Claude Huriez, Lille, Cedex
  - Hospital Haut Leveque, Pessac, Cedex
  - Hospital Cavale Blanche, Brest
- Germany (3):
  - Universitaetsklinikum Dresden, Dresden
  - University Hospital Greifswald, Greifswald
  - Universitaetsklinikum Heidelberg, Heidelberg
- Israel (3):
  - Pulmonology Department Rambam Medical Center, Haifa
  - Lady Davis Carmel Medical Centre, Haifa
  - Pulmonary institute, Ramat Gan
- Azienda Ospedaliera Universitaria, Naples, Italy
- VUMC, Amsterdam, Netherlands
- Hospital de Santa Marta, Lisbon, Portugal
- Spain (2):
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
- Lund University Hospital, Lund, Sweden
- Royal Free Hospital NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Lachant D, Raina A, Krishnan M, Sood N, Balasubramanian V, Barbera JA, Kiely DG, Lee D, Wu B, Hwang S, Seaman S, Broderick M, Elwing J. Efficacy and Safety of Oral Treprostinil in Patients with Pulmonary Arterial Hypertension on Background Monotherapy or Dual Therapy. Adv Ther. 2026 Feb 2. doi: 10.1007/s12325-026-03497-4. Online ahead of print. PMID 41627369
- [Derived] Richter MJ, Schermuly R, Seeger W, Rao Y, Ghofrani HA, Gall H. Relevance of angiopoietin-2 and soluble P-selectin levels in patients with pulmonary arterial hypertension receiving combination therapy with oral treprostinil: a FREEDOM-C2 biomarker substudy. Pulm Circ. 2016 Dec;6(4):516-523. doi: 10.1086/688671. PMID 28090293
- [Derived] Tapson VF, Jing ZC, Xu KF, Pan L, Feldman J, Kiely DG, Kotlyar E, McSwain CS, Laliberte K, Arneson C, Rubin LJ; FREEDOM-C2 Study Team. Oral treprostinil for the treatment of pulmonary arterial hypertension in patients receiving background endothelin receptor antagonist and phosphodiesterase type 5 inhibitor therapy (the FREEDOM-C2 study): a randomized controlled trial. Chest. 2013 Sep;144(3):952-958. doi: 10.1378/chest.12-2875. PMID 23669822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was June 2009 to July 2011. Sites were located in North America, Europe and Asia.
Pre-assignment Details: The 310 subjects who received a dose of study drug are presented here.
Period: Overall Study
Arm/Group | UT-15C SR | Placebo
Started | 157 | 153
Completed | 132 | 138
Not Completed | 25 | 15
Not completed — Adverse Event | 18 | 5
Not completed — Clinical Worsening | 4 | 4
Not completed — Death | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UT-15C SR | Placebo | Total
Number analyzed (Participants) | 157 | 153 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 122 | 241
  >=65 years | 38 | 31 | 69
Age Continuous [Mean (Full Range); unit: years] | 51.5 (15) [18 to 76] | 50.4 (14.5) [20 to 75] | 51.0 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 122 | 241
  Male | 38 | 31 | 69
PAH Etiology [Number; unit: participants]
  Idiopathic or familial | 104 | 99 | 203
  Collagen vascular disease | 48 | 49 | 97
  HIV infection | 2 | 4 | 6
  Repaired congenital heart disease | 3 | 1 | 4
World Health Organization (WHO) Functional Class [Number; unit: Participants] — Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
  Participants
    Class II | 43 | 37 | 80
    Class III | 110 | 115 | 225
    Class IV | 3 | 0 | 3
    Unknown | 1 | 1 | 2
Baseline Six-minute walk distance [Mean (Standard Deviation); unit: meters] | 329.4 (69.2) | 336.8 (63.5) | 333 (66.4)
Background PAH therapy [Number; unit: participants] — Eligible subjects were receiving background PAH therapy of either a phosphodiesterase-5 inhibitor (PDE-5i) and/or endothelin receptor antagonist (ERA)
  participants
    PDE-5i | 67 | 65 | 132
    ERA | 25 | 28 | 53
    PDE-5i + ERA | 65 | 60 | 125
Time since PAH diagnosis [Mean (Standard Deviation); unit: years] | 2.5 (2.6) | 3.3 (4.1) | 2.9 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: 6-minute Walk Distance (6MWD)
Description: Placebo-corrected change in 6MWD from Baseline to Week 16, correlates with the current clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The 6MWD was to be assessed between 3 and 6 hours after the morning dose of study drug and background therapy(ies).
Time Frame: Baseline and 16 weeks
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- UT-15C SR: At Week 16, the mean(SD) dose of UT-15C was 3.1mg (1.9).
- Placebo: At Week 16, the mean(SD) dose of placebo was 6.1mg (3.6).
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 157 | 153
meters
  Week 16 Values | 370 [292 to 419] | 365 [300 to 405]
  Change from Baseline | 15 [-12 to 55] | 11 [-14 to 39]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Using an allocation ratio of 1:1 between UT-15C SR and placebo, a fixed sample size of approximately 266 subjects would provide at least 90% power at a significance level of 0.05 (two-sided hypothesis) to detect a 30 meter between-treatment difference in the change from Baseline in distance traversed during the 6-Minute Walk, assuming a standard deviation of 75 meters. A total sample size of approximately 300 subjects was determined to account for discontinuations during the enrollment period; Test type: Superiority or Other; p = 0.089, non-parametric ANCOVA; Hodges-Lehmann (H-L) = 10.0, 95% CI 2-sided [-2.0 to 22.0]

2. Secondary Outcome: Clinical Worsening Assessment
Description: Definition of clinical worsening included patients who met at least one of the following criteria during the 16 weeks of study:
  1. Death (all causes excluding accident)
  2. Transplantation
  3. Atrial septostomy
  4. Hospitalization as a result of right heart failure
  5. Greater than or equal to a 20% decrease in 6MWD from Baseline (or too ill to walk) AND addition of an inhaled prostacyclin analogue, ERA, or PDE-5i
  6. Initiation of parenteral prostacyclin therapy (i.e., epoprostenol, iloprost, or treprostinil) for the treatment of PAH
Time Frame: Baseline and 16 Weeks
Population: Intention to treat analysis
Measure: Number; unit: number of clinical worsening events
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 157 | 153
number of clinical worsening events | 11 | 10
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact

3. Secondary Outcome: Borg Dyspnea Score
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the six-minute walk test (6MWT). The Borg dyspnea score was assessed immediately following the 6MWT. Scores ranged from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced).
Time Frame: Baseline and 16 Weeks
Population: All subjects with a Baseline Borg Score were included in the analysis. One subject in the placebo group did not have a Baseline Borg Score recorded.
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 157 | 152
score
  Week 16 Value | 3.0 (2.47) [2.0 to 5.0] | 4.0 (2.05) [2.0 to 5.0]
  Change from Baseline | 0 [-1.0 to 1.0] | 0 [-1.0 to 1.0]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.22, Wilcoxon rank sum test; Hodges-Lehmann (H-L) Estimate = 0.0, 95% CI 2-sided [-1.0 to 0.0]

4. Secondary Outcome: World Health Organization (WHO) Functional Class
Description: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
Time Frame: Baseline and 16 Weeks
Population: Subjects with a WHO functional class assessment at Week 16
Measure: Number; unit: participants
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 131 | 136
participants
  WHO Class I | 1 | 3
  WHO Class II | 58 | 47
  WHO Class III | 70 | 83
  WHO Class IV | 2 | 3
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.43, Wilcoxon rank sum test — Imputation strategies were implemented for the 26 UT-15C subjects and 17 placebo subjects without values reported at Week 16; Hodges-Lehmann (H-L) estimate = 0.0, 95% CI 2-sided [0.0 to 0.0]

5. Secondary Outcome: Symptoms of PAH
Description: Symptoms of PAH including fatigue, dyspnea, edema, dizziness, syncope, chest pain and orthopnea were assessed by the physician at Baseline and Week 16. Severity grade values (i.e., 0, 1, 2 or 3) for each symptom were provided each subject. A severity of 0 indicated no symptoms, the maximum severity was 3, indicating severe symptoms. Mean change in symptom severity from Baseline to Week 16 is described.
Time Frame: Baseline and 16 Weeks
Population: Subjects without Baseline assessments of PAH symptoms were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 156 | 150
units on a scale
  Change in Fatigue Symptoms | 0.0 (0.9) | 0.0 (1.0)
  Change in Dyspnea Symptoms | -0.1 (0.9) | -0.2 (0.9)
  Change in Edema Symptoms | 0.0 (1.0) | 0.0 (0.9)
  Change in Dizziness Symptoms | 0.1 (1.0) | 0.0 (1.0)
  Change in Syncope Symptoms | 0.2 (0.8) | 0.2 (0.7)
  Change in Chest Pain Symptoms | 0.1 (1.0) | 0.1 (1.0)
  Change in Orthopnea Symptoms | 0.2 (1.0) | 0.1 (0.9)

6. Secondary Outcome: Dyspnea Fatigue Index
Description: The dyspnea-fatigue index was assessed at Baseline and Week 16. Each of the three components of the dyspnea-fatigue index were rated on a scale 0 to 4, with 0 being the worst condition and 4 being the best condition for each component. The dyspnea-fatigue index is computed by summing the three component scores.
Time Frame: Baseline and 16 Weeks
Population: Subjects without a Dyspnea Fatigue Index score at Baseline were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 154 | 149
units on a scale | 5.7 (2.6) | 6.0 (2.5)
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.30, Wilcoxon rank sum test; Hodges-Lehmann (H-L) estimate = 0.0, 95% CI 2-sided [0.0 to 1.0]

7. Secondary Outcome: N-terminal proBNP (NT-proBNP)
Description: Serum N-terminal pro-BNP concentration was assessed at Baseline and Week 16.
Time Frame: Baseline and 16 Weeks
Population: Subjects who were missing Week 16 samples were not included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 120 | 135
pg/mL
  Week 16 Value | 1310 (1663) | 1627 (2401)
  Change from Baseline | 135 (913) | 136 (1242)

8. Secondary Outcome: Quality of Life (QoL) Assessment: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR)
Description: Change in CAMPHOR Scores from Baseline to Week 16. The CAMPHOR is a health related quality of life instrument validated for pulmonary hypertension that assesses impairment (symptoms), disability (activities) and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 0-25; high scores indicate more symptoms), Activity (Score 0-30; low score indicates good functioning)and Quality of Life (0-25; high scores indicate poor QoL). The sum of these scores equates to the Total score (0-80). In the CAMPHOR scores, lower scores indicate improvements.
Time Frame: Baseline and 16 Weeks
Population: Subjects in countries where the CAMPHOR has not been validated in the local language were not included in these analyses. Additionally, only subjects with completed questionnaires at Baseline and Week 16 were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 102 | 85
units on a scale
  Symptom Score | 10.0 [6.0 to 16.0] | 9.0 [4.0 to 14.0]
  Activity Score | 10.0 [7.0 to 14.0] | 10.0 [6.0 to 13.0]
  Quality of Life Score | 9.0 [4.0 to 15.0] | 5.0 [1.5 to 13.0]
  Total Score | 28.0 [19.0 to 43.0] | 24.5 [12.0 to 40.5]

9. Post Hoc Outcome: 6-minute Walk Distance by PAH Etiology: Idiopathic PAH (IPAH) / Heritable PAH(HPAH)
Description: Covariate analysis of change in 6MWD by PAH etiology, specifically idiopathic or heritable PAH
Time Frame: Baseline and 16 Weeks
Population: Subjects with IPAH/HPAH
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 104 | 99
meters | 21.5 [-0.5 to 64.5] | 13 [-14 to 39]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.058, ANCOVA; Hodges-Lehman Estimate = 14.0, 95% CI 2-sided [0.0 to 28.0]

10. Post Hoc Outcome: 6-minute Walk Distance by Background PAH Therapy: PDE-5i Only
Time Frame: 16 weeks
Population: Subjects receiving only a PDE-5i at Baseline
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 67 | 65
meters | 30 [4 to 55] | 14 [-7 to 39]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.054, ANCOVA; Hodges-Lehmann Estimate = 15.0, 95% CI 2-sided [-1.0 to 29.0]

11. Post Hoc Outcome: 6-minute Walk Test by Background PAH Therapy: ERA Only
Time Frame: Baseline and 16 weeks
Population: Subjects who were only receiving an ERA at Baseline
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 25 | 28
meters | -5 [-43.0 to 42.0] | -2.5 [-49.0 to 30.0]

12. Post Hoc Outcome: 6-minute Walk Test by Background PAH Therapy: ERA + PDE-5i
Time Frame: 16 weeks
Population: Subjects receiving both an ERA and a PDE-5i at Baseline.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 65 | 60
meters | 14.0 [-17 to 59] | 15.5 [-14.5 to 39]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.674, ANCOVA; Hodges-Lehman Estimate = 4.0, 95% CI 2-sided [-16.0 to 24.0]

13. Post Hoc Outcome: 6-minute Walk Distance by Time to PAH Diagnosis: 0 - 0.9 Years
Time Frame: Baseline and 16 weeks
Population: Subjects who have been diagnosed with PAH between 0 to 0.9 years prior to Baseline.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 40 | 38
meters | 21.5 [-12.5 to 50.5] | -6.0 [-63.0 to 26.0]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.059, ANCOVA; Hodges-Lehmann Estimate = 28.0, 95% CI 2-sided [1.0 to 59.0]

14. Post Hoc Outcome: 6-minute Walk Distance by Time Since PAH Diagnosis: 0.9 - 1.74 Years
Time Frame: 16 Weeks
Population: Subjects who had been diagnosed with PAH between 0.9 and 1.74 years prior to Baseline.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 40 | 37
meters | 20.1 [1.0 to 61.0] | 13.0 [-2.0 to 45.0]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.22, ANCOVA; Hodges-Lehmann Estimate = 10.0, 95% CI 2-sided [-10.0 to 31.0]

15. Post Hoc Outcome: 6-minute Walk Distance by Years Since PAH Diagnosis: 1.8 - 3.5 Years
Time Frame: Baseline and 16 weeks
Population: Subjects who were diagnosed with PAH between 1.8 and 3.5 years prior to Baseline.
Measure: Median (Inter-Quartile Range); unit: meter
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 40 | 37
meter | 15.5 [-16.0 to 51.5] | 4.0 [-14.0 to 42.0]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.99, ANCOVA; Hodges-Lehmann Estimate = 3.0, 95% CI 2-sided [-23.0 to 28.0]

16. Post Hoc Outcome: 6-minute Walk Distance by Time Since PAH Diagnosis: 3.6 - 26.4 Years
Time Frame: Baseline and 16 weeks
Population: Subjects who had been diagnosed with PAH for 3.6 to 26.4 years prior to Baseline.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | UT-15C SR | Placebo
Number analyzed (Participants) | 37 | 41
meters | 14.0 [-23.0 to 59.0] | 16.0 [-5.0 to 36.0]
Statistical Analysis 1: Comparison: UT-15C SR vs Placebo; Test type: Superiority or Other; p = 0.84, ANCOVA; Hodges-Lehmann Estimate = -2.0, 95% CI [-25.0 to 22.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 16 week study.
Groups:
- UT-15C SR: At Week 16, the mean(SD) dose of UT-15C was 3.1 (1.9).
- Placebo: At Week 16, the mean(SD) dose of placebo was 6.1 (3.6).
Arm/Group | UT-15C SR | Placebo
Serious Adverse Events (participants affected / at risk) | 23/157 | 23/153
Other Adverse Events (participants affected / at risk) | 157/157 | 136/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR (N=157) | Placebo (N=153)
Right ventricular failure (Cardiac disorders) | 5 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hypervolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2)
Peripheral edema (General disorders) | 0 (0) | 1 (1)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Hepatic ischemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR (N=157) | Placebo (N=153)
Headache (Nervous system disorders) | 112 (145) | 61 (69)
Diarrhea (Gastrointestinal disorders) | 87 (105) | 38 (42)
Nausea (Gastrointestinal disorders) | 73 (77) | 34 (35)
Flushing (Vascular disorders) | 55 (64) | 16 (18)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 39 (39) | 10 (10)
Vomiting (Gastrointestinal disorders) | 33 (38) | 16 (20)
Dizziness (Nervous system disorders) | 30 (36) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (29) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 10 (15)
Fatigue (General disorders) | 23 (25) | 16 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (18) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 13 (13)
Peripheral edema (General disorders) | 17 (18) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 12 (13) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (12) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 11 (12) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 25 (28)
Chest Pain (General disorders) | 9 (9) | 10 (11)
Palpitations (Cardiac disorders) | 6 (6) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.